CLINICAL TRIAL: NCT01165736
Title: An Exploratory, Open Label, Randomized, Parallel Group Study To Investigate The Pharmacokinetics Of Single Intravenous And Oral Micro Doses Of PF-05186462, PF-05089771, PF-05241328 And PF-05150122 In Healthy Male Subjects
Brief Title: To Calculate the Pharmacokinetics (Concentration of Compound in and Rate of Excretion From the Blood) Following a Very Low Dose of Compound Which Will Not Have Any Pharmacological Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B3071001
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: pharmacokinetics; safety; tolerability; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — PF-05089771

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Intravenous: PF-05186462 (Active Comparator)
  Interventions: Drug: PF-05186462
- Oral: PF-05186462 (Active Comparator)
  Interventions: Drug: PF-05186462
- Intravenous: PF-05089771 (Active Comparator)
  Interventions: Drug: PF-05089771
- Oral: PF-05089771 (Active Comparator)
  Interventions: Drug: PF-05089771
- Intravenous: PF-05150122 (Active Comparator)
  Interventions: Drug: PF-05150122
- Oral: PF-05150122 (Active Comparator)
  Interventions: Drug: PF-05150122
- Intravenous: PF-05241328 (Active Comparator)
  Interventions: Drug: PF-05241328
- Oral: PF-05241328 (Active Comparator)
  Interventions: Drug: PF-05241328

INTERVENTIONS:
Drug: PF-05186462 — single intravenous infusion of 100 microgram
  Arms: Intravenous: PF-05186462
Drug: PF-05186462 — single oral administration of 100 microgram
  Arms: Oral: PF-05186462
Drug: PF-05089771 — single intravenous infusion of 100 microgram of PF-05089771
  Arms: Intravenous: PF-05089771
Drug: PF-05089771 — single oral administration of 100 microgram PF-05089771
  Arms: Oral: PF-05089771
Drug: PF-05150122 — single intravenous administration of 100 microgram PF-05150122
  Arms: Intravenous: PF-05150122
Drug: PF-05150122 — single oral administration of 100 microgram PF-05150122
  Arms: Oral: PF-05150122
Drug: PF-05241328 — single intravenous infusion of 100 microgram PF-05241328
  Arms: Intravenous: PF-05241328
Drug: PF-05241328 — single oral administration 100 microgram PF-05241328
  Arms: Oral: PF-05241328

SUMMARY:
The purpose of this study is to calculate the pharmacokinetics (concentration of compound in and rate of excretion from the blood) following a very low dose of compound which will not have any pharmacological activity and to monitor for the safety and tolerability of each of the compounds in the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects between the ages of 18 and 50 years inclusive. (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests)
* Body Mass Index (BMI) of 17.5 to 30.5kg/m2l and a total body weight of between 50 and 100kg inclusive.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, genitourinary, psychiatric, neurologic or allergic disease (including drug allergies, but excluding untreated, symptomatic, seasonal allergies at time of dosing)
* History of febrile illness within 5 days prior to the first dose a positive urine drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (heart rate, blood pressure, QTcF, clinical chemistry) | up to 3 days post dose
pharmacokinetics of each of the four compounds measuring Clearance, volume of distribution, elimination half life and area under the effect curve | up to 3 days post dose

SECONDARY OUTCOMES:
safety and tolerability of each of the four compounds (heart rate, blood pressure, QTcF, clinical chemistry) | up to 3 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Edinburgh, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3071001&StudyName=To%20calculate%20the%20pharmacokinetics%20%28concentration%20of%20compound%20in%20and%20rate%20of%20excretion%20from%20the%20blood%29%20following%20a%20very%20low%20dose%20of